CLINICAL TRIAL: NCT06328101
Title: A Multicenter, Retrospective Study on Autoimmune Pancreatitis, Pancreatic and Extrapancreatic cAnceR (AiPPEAR)
Brief Title: Autoimmune Pancreatitis, Pancreatic and Extrapancreatic cAnceR (AiPPEAR)
Acronym: AiPPEAR
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Collaborators: University Medical Centre Maribor (Other); Aalborg University Hospital (Other); University Hospital Munich (Other); Tartu University Hospital (Other); University Hospital in Halle (Other)
Responsible Party: Principal Investigator, Christoph Ammer-Herrmenau, Medical Doctor, University Medical Center Goettingen
Other Study IDs: 2023-02558
Record Dates: First submitted 2024-02-15; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Autoimmune Pancreatitis Type 1; Autoimmune Pancreatitis Type 2
Keywords: autoimmune pancreatitis; cancer; risk; pancreatic cancer; hepatobiliary cancer
MeSH Terms: conditions — Autoimmune Pancreatitis; Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AIP_mlg: Autoimmune pancreatitis patients with cancer
- AIP_nomlg: Autoimmune pancreatiits patients without cancer
- general population: Cancer Incidence in Five Continents Volume XI" (CI5XI) registry patients used to determine expected cancer incidence and calculate SIR

SUMMARY:
The goal of this observational, retrospective study is to learn about cancer risk in autoimmune pancreatitis (AIP) patients. The main questions it aims to answer are:

* Do patients with AIP have higher incidence of cancer in comparison to general population?
* What is the overall prevalence of cancer in AIP patients?
* What are the characteristics of AIP patients associated with the incidence of cancer?

DETAILED DESCRIPTION:
Autoimmune pancreatitis (AIP) is a relapsing form of pancreatitis, comprising two histological entities with differing clinical, serological, and prognostic characteristics. Type 1 AIP is a pancreatic manifestation of IgG4-related disease, while type 2 AIP is an isolated pancreatic disorder strongly associated with the simultaneous occurrence of inflammatory bowel disease (IBD). AIP patients, particularly type 1, face a risk of relapse and may develop exocrine and endocrine pancreatic insufficiency. While it's widely acknowledged that chronic pancreatitis increases the risk of pancreatic cancer, the association between AIP and pancreatic cancer remains more controversial. AIP can imitate pancreatic cancer, and coincidence has been reported. Retrospective data from Japan suggested a high risk of pancreatic cancer and bile duct cancer in patients with AIP. However, there is a paucity of specific data on the relationship between AIP and pancreatic cancer. Japanese studies have suggested a higher incidence of extrapancreatic cancer in AIP patients compared to the general population. German single-center data support this claim. The most frequently reported cancers include lung, gastric, and prostate cancer, constituting approximately 50% of all cancers detected at or after the diagnosis of AIP. However, the time span of both AIP and cancer was not defined and might have introduced bias. Available data need to be interpreted with caution as no studies have yet compared the incidence of the most common cancers in AIP patients directly to age-grouped and gender-matched controls in the general population.

To address this lack of knowledge a worldwide, multicenter, retrospective cohort study of AIP patients is initiated founded in the Pancreas2000 framework. With this trial cancer incidence and prevalence will be assessed for AIP patients and compared to age-matched controls.

The trial is based on a REDCap questionnaire containing following information.

1. Demographic details Month and year of birth Survival status month and year of death, if applicable Gender (Male, Female) Ethnicity (Caucasian, Hispanic, African, Asian, Arabic, Other, Unknown) Weight and height for the purpose of calculating body mass index Tobacco status (Current, Former, Never) incl. "smoking pack-years" if applicable Alcohol consumption (Current daily, current occasionally, Former, Never, Not available) History of other autoimmune diseases (not IgG4-related) (No, Sjögren's' syndrome, Rheumatoid arthritis, Sarcoidosis, Autoimmune thyroiditis (NOT IgG4 related), Other) History of inflammatory bowel disease (Yes, No, Unknown) Family history of cancer (Yes, No, Unknown)
2. AIP characteristics Month and year of diagnosis AIP The classification system used for original diagnosis (ICDC, HISORT, Asian, Unify) ICDC diagnosis type (Type 1, Type 2, Not otherwise specified (NOS) AIP) ICDC diagnosis level (Definite, Probable) ICDC parameters fulfilled for diagnosis (Histology, Serum IgG4, Imaging, Improvement after steroid treatment, Other organ involvement) Serum IgG4 (1-2 over upper limit, >2 over the upper limit, >4 over the upper limit) Imaging (Focal enlargement, Whole organ enlargement (sausage-like), Other) Other organ involvement (Salivary/lacrymal glands, Retroperitoneum/ kidneys, Bile ducts/liver, Musculoskeletal system, Gastrointestinal tract: Intestines, colon, esophagus, Vasculitis (e.g., aortitis), Enlarged lymph nodes, IBD) Presenting symptoms of AIP (None, Jaundice, Acute pancreatitis, Weight loss, Abdominal pain, New onset of diabetes) Medical treatment for AIP (Prednisone, Rituximab, Azathioprine, 6-mercaptopurine, Methotrexate, Mycophenolate mofetil, other) Interventional treatment for AIP (Partial pancreatectomy, Biliary stent placement, Other) AIP relapse (No relapse, 1-2 relapse(s), 3-4 relapses, >5 relapses, Unknown) AIP-related complications (No, Diabetes mellitus, Pancreatic exocrine insufficiency, Other) Month and year of last contact
3. Cancer Diagnosis Month and year of diagnosis of cancer Number of cancer diseases (1,2,3,4) Cancer type (list according to the World Health Organization) Cancer-related death (yes, no) In case of more than one cancer, specifically which cancer caused death

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AIP after 2005, including type 1, type 2, and not-otherwise-specified (NOS) AIP, regardless of the diagnostic criteria used.

Exclusion Criteria:

* Patients younger than 18 years at last contact
* Patients with less than 12 months of follow up after diagnosis
* Patients with immune checkpoint inhibitor-induced pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary centers specializing in the treatment of pancreatitis worldwide will be invited to participate in the study. Patients with AIP will be identified locally, and information for characterization of risk factors, AIP, and cancer will be retrospectively extracted from the medical files. The core group comprises six centers from Denmark, Germany, Slovenia, and Estonia.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Standardized incidence ratio (SIR) of first invasive cancer | up to 20 years
  The standardized incidence ratio (SIR) of the first invasive cancer occurring after the diagnosis of AIP compared to age-grouped and gender-matched controls in the general population. We will count the incidence of invasive cancer in AIP patients (yes/no).

SECONDARY OUTCOMES:
The prevalence of cancer diagnoses 12 months prior to AIP diagnosis | 12 months prior to AIP diagnosis
  We will count if there is a previous cancer diagnosis (yes/no) and from medical records (ICD code according to cancer registry) 12 moths prior to AIP diagnosis and determine prevalence in %
Risk factor associated with cancer diagnosis. | up to 20 years
  For every case other possible risk factor for cancer will be assesed such as the gender (female, male), the body mass index (BMI), the type of AIP (type 1, type 2), smoking, diabetes mellitus after diagnosis of AIP , Elevate IgG4 levels at diagnosis, maintainance treatmet, other organ involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie Siggaard Knoph, MD, Principal Investigator — Univesity Hospital Alborg; Julian Cardinal von Widdern, MD, Principal Investigator — University Hospital Halle (Saale); Karri Kasse, MD, Principal Investigator — Tartu University Hospital; Ivonne Regel, PhD, Study Chair — University Hospital of Munich (LMU); Jonas Rosendahl, MD, PhD, Study Chair — University Hospital Halle (Saale)

IPD SHARING:
Plan to Share IPD: No
IPD will be available only to core group, not other researches. Core group retains right to perform post-hoc analyses, these proposals will be reviewed and granted by the steering committee.

REFERENCES:
- [Background] Lohr JM, Beuers U, Vujasinovic M, Alvaro D, Frokjaer JB, Buttgereit F, Capurso G, Culver EL, de-Madaria E, Della-Torre E, Detlefsen S, Dominguez-Munoz E, Czubkowski P, Ewald N, Frulloni L, Gubergrits N, Duman DG, Hackert T, Iglesias-Garcia J, Kartalis N, Laghi A, Lammert F, Lindgren F, Okhlobystin A, Oracz G, Parniczky A, Mucelli RMP, Rebours V, Rosendahl J, Schleinitz N, Schneider A, van Bommel EF, Verbeke CS, Vullierme MP, Witt H; UEG guideline working group. European Guideline on IgG4-related digestive disease - UEG and SGF evidence-based recommendations. United European Gastroenterol J. 2020 Jul;8(6):637-666. doi: 10.1177/2050640620934911. Epub 2020 Jun 18. PMID 32552502
- [Background] Shimosegawa T, Chari ST, Frulloni L, Kamisawa T, Kawa S, Mino-Kenudson M, Kim MH, Kloppel G, Lerch MM, Lohr M, Notohara K, Okazaki K, Schneider A, Zhang L; International Association of Pancreatology. International consensus diagnostic criteria for autoimmune pancreatitis: guidelines of the International Association of Pancreatology. Pancreas. 2011 Apr;40(3):352-8. doi: 10.1097/MPA.0b013e3182142fd2. PMID 21412117
- [Background] Nikolic S, Lanzillotta M, Panic N, Brismar TB, Moro CF, Capurso G, Della Torre E, Lohr JM, Vujasinovic M. Unraveling the relationship between autoimmune pancreatitis type 2 and inflammatory bowel disease: Results from two centers and systematic review of the literature. United European Gastroenterol J. 2022 Jun;10(5):496-506. doi: 10.1002/ueg2.12237. Epub 2022 May 8. PMID 35526270
- [Background] Lee HW, Moon SH, Kim MH, Cho DH, Jun JH, Nam K, Song TJ, Park DH, Lee SS, Seo DW, Lee SK. Relapse rate and predictors of relapse in a large single center cohort of type 1 autoimmune pancreatitis: long-term follow-up results after steroid therapy with short-duration maintenance treatment. J Gastroenterol. 2018 Aug;53(8):967-977. doi: 10.1007/s00535-018-1434-6. Epub 2018 Jan 23. PMID 29362937
- [Background] Lanzillotta M, Tacelli M, Falconi M, Arcidiacono PG, Capurso G, Della-Torre E. Incidence of endocrine and exocrine insufficiency in patients with autoimmune pancreatitis at diagnosis and after treatment: a systematic review and meta-analysis. Eur J Intern Med. 2022 Jun;100:83-93. doi: 10.1016/j.ejim.2022.03.014. Epub 2022 Mar 30. PMID 35367110
- [Background] Nikolic S, Maisonneuve P, Dahlman I, Lohr JM, Vujasinovic M. Exocrine and Endocrine Insufficiency in Autoimmune Pancreatitis: A Matter of Treatment or Time? J Clin Med. 2022 Jun 28;11(13):3724. doi: 10.3390/jcm11133724. PMID 35807009
- [Background] Lowenfels AB, Maisonneuve P, Cavallini G, Ammann RW, Lankisch PG, Andersen JR, Dimagno EP, Andren-Sandberg A, Domellof L. Pancreatitis and the risk of pancreatic cancer. International Pancreatitis Study Group. N Engl J Med. 1993 May 20;328(20):1433-7. doi: 10.1056/NEJM199305203282001. PMID 8479461
- [Background] Kurita Y, Kubota K, Fujita Y, Tsujino S, Sekino Y, Kasuga N, Iwasaki A, Iwase M, Izuka T, Kagawa K, Tanida E, Yagi S, Hasegawa S, Sato T, Hosono K, Kobayashi N, Ichikawa Y, Nakajima A, Endo I. IgG4-related pancreatobiliary diseases could be associated with onset of pancreatobiliary cancer: A multicenter cohort study. J Hepatobiliary Pancreat Sci. 2024 Mar;31(3):173-182. doi: 10.1002/jhbp.1404. Epub 2023 Dec 20. PMID 38124014
- [Background] Shiokawa M, Kodama Y, Yoshimura K, Kawanami C, Mimura J, Yamashita Y, Asada M, Kikuyama M, Okabe Y, Inokuma T, Ohana M, Kokuryu H, Takeda K, Tsuji Y, Minami R, Sakuma Y, Kuriyama K, Ota Y, Tanabe W, Maruno T, Kurita A, Sawai Y, Uza N, Watanabe T, Haga H, Chiba T. Risk of cancer in patients with autoimmune pancreatitis. Am J Gastroenterol. 2013 Apr;108(4):610-7. doi: 10.1038/ajg.2012.465. Epub 2013 Jan 15. PMID 23318486
- [Background] Schneider A, Hirth M, Munch M, Weiss C, Lohr JM, Ebert MP, Pfutzer RH. Risk of Cancer in Patients with Autoimmune Pancreatitis: A Single-Center Experience from Germany. Digestion. 2017;95(2):172-180. doi: 10.1159/000455963. Epub 2017 Feb 23. PMID 28226313
- [Derived] Cardinal von Widdern J, Knoph CS, Kase K, Regel I, Rosendahl J, Ammer-Hermenau C, Nikolic S. Autoimmune pancreatitis, pancreatic and extrapancreatic cancer (AIPPEAR): a multicentre, retrospective study protocol. BMJ Open. 2025 Feb 16;15(2):e086824. doi: 10.1136/bmjopen-2024-086824. PMID 39956600